CLINICAL TRIAL: NCT04346654
Title: A Phase II, Randomized (1:1) Open Label Study to Assess the Efficacy and Safety of Eltrombopag in Combination With Dexamethasone Compared to Dexamethasone, as First-line Treatment in Adult Patients With Newly Diagnosed Immune Thrombocytopenia
Brief Title: A Study to Assess Efficacy and Safety of Eltrombopag in Combination With a Short Course of Dexamethasone in Patients With Newly Diagnosed ITP
Acronym: XPAG-ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETB115JDE01; 2019-002658-21 (EudraCT Number)
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: ITP; Eltrombopag; Dexamethasone; Sustained response off treatment; TFR; Adult; ETB115; Platelets; Thrombocytopenic; Thrombopoietin receptor Agonist; Newly-diagnosed; Blood bleeding disorder
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag + Dexamethasone (Experimental): Patients were treated with eltrombopag in combination with a standard high-dose dexamethasone (1 cycle: 40 mg once daily (QD) from day 1-4) to induce sustained response off treatment.
  Interventions: Drug: Eltrombopag; Drug: Dexamethasone
- Dexamethasone (Active Comparator): Patients were treated with a standard high-dose dexamethasone (1-3 cycles: 40 mg QD day 1-4 at 4 weeks intervals (or at 14-28 days intervals if needed) to induce sustained response off treatment.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag is for oral use and comes in 25, 50 and 75 mg tablets. Prescribed dose is taken once daily.
  Other Names: ETB115
  Arms: Eltrombopag + Dexamethasone
Drug: Dexamethasone — Dexamethasone is for oral use and comes in 8 mg tablets. Prescribed dose is taken once daily.

SUMMARY:
The purpose of this study was to compare the ability of eltrombopag in combination with a short course of high-dose dexamethasone to induce sustained response off treatment in patients with newly-diagnosed ITP versus 1-3 cycles of dexamethasone monotherapy.

The unmet clinical need and the potential for eltrombopag when added to steroids to improve the treatment outcome and the potential to induce sustained response off treatment serve as the basis for clinical investigation of eltrombopag in first-line ITP.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, 1:1 randomized, open-label study that compared the efficacy and safety of eltrombopag in combination with a short course of high-dose dexamethasone to 1-3 cycles of high-dose dexamethasone monotherapy, as first-line treatment in adult patients with newly diagnosed ITP.

Adult patients with newly diagnosed ITP who had platelet counts < 30 × 10^9/L and required treatment were screened, and if eligible, were randomized to either Arm A (eltrombopag in combination with a short course of dexamethasone) or Arm B (1-3 cycles of dexamethasone monotherapy).

The study was conducted in the following periods:

Screening Period: Patients were screened for 14 days based on the inclusion and exclusion criteria.

Treatment Period: Arm A: Patients were treated for 26 weeks during the treatment period. Patients who reached platelet counts ≥ 30 × 10^9/L and maintained counts ≥ 30 × 10^9/L during the tapering phase were eligible for treatment discontinuation. Duration of tapering before treatment discontinuation at Week 26 was 6 weeks. Arm B: Patients were treated up to 12 weeks during the treatment period. Patients who reached platelet counts ≥ 30 × 10^9/L and maintained counts ≥ 30 × 10^9/L after 1-3 cycles of dexamethasone treatment were eligible for treatment discontinuation. Patients with platelet counts < 30 × 10^9/L after 3 cycles of dexamethasone treatment were offered a course of eltrombopag treatment within the study and were discontinued from study at week 52.

Observation period: After completion of the treatment period, all patients were observed for sustained response off treatment until week 52. Only patients with sustained response at week 52 were followed for another 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Men and women ≥ 18 years of age
* Newly diagnosed with primary ITP (time from diagnosis within 3 months)
* Platelet count < 30 × 109/L at screening and a need for treatment (per physician's discretion) Note: If pre-treatment is necessary, platelet count data performed directly before pre-treatment (can be used for study inclusion (screening value). Treatment-naïve patients will be included based on their platelet counts performed at screening

Exclusion Criteria:

* Previous history of treatment for ITP, except any ITP-directed therapy for a maximum of 3 days within 7 days before randomization
* Patients with diagnosis of secondary thrombocytopenia
* Patients who have life threatening bleeding complications per physician´s discretion
* Patients with a history of thromboembolic events in the 6 months preceding enrollment or known risk factors for thromboembolism
* Serum creatinine > 1.5 mg/dL
* Total bilirubin (TBIL) > 1.5 × upper limit of normal (ULN)
* Aspartate transaminase (AST) > 3.0 × ULN
* Alanine transaminase (ALT) > 3.0 × ULN
* Patients who are human immune deficiency virus (HIV),hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg) positive
* Patients with hepatic impairment (Child-Pugh score > 5)
* Patients with known active or uncontrolled infections not responding to appropriate therapy
* History of current diagnosis of cardiac disease or impaired cardiac function denoted
* Patients who have active malignancy
* Patients with evidence of current alcohol/drug abuse
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures
* Female subjects who are nursing or pregnant (positive serum or urine B-human chorionic gonadotrophin (B-hCG) pregnancy test) at screening or pre-dose on Day 1
* Women of child-bearing potential and males unwilling to use adequate contraception during the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaacueticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Kronach

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 25 centers in Germany.
Pre-assignment Details: Participants had to abstain from using investigational/marketed drugs and taking herbal supplements prior to taking the first dose of study treatment.
Period: Overall Study
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Started | 13 | 13
Randomized, Not Treated | 1 | 0
Completed (Completed = Completed after Week 52) | 8 | 10
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Non-response | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (14.5) | 45.3 (14.3) | 53.0 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 12 | 12 | 24
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Sustained Response Off Treatment at 52 Weeks
Description: Sustained response off treatment at 52 weeks is defined as maintenance of platelet count ≥ 30 × 10^9/L after treatment discontinuation until Week 52 in the absence of bleeding events ≥ Grade II or use of any rescue medication at all visits until Week 52. Bleeding events ≥ Grade II are assessed by the modified World Health Organization (WHO) Bleeding Scale; Bleeding is graded based on a 1-4 scale (1=minor bleeding to 4=severe bleeding). Characteristics of bleeding events ≥ Grade II include: epistaxis ≥30 minutes, large purpura, joint bleeding, melanotic stool, hematemesis, gross hematuria, abnormal vaginal bleeding, hemoptysis, Visible blood in body cavity fluid, retinal bleeding, bleeding at invasive sites, bleeding requiring transfusion, bleeding associated with moderate or severe hemodynamic instability, fatal bleeding, CNS bleeding.
Time Frame: Study treatment discontinuation until week 52
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Participants | 2 | 2
Statistical Analysis 1: Comparison: Eltrombopag + Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.5133, Regression, Logistic

2. Secondary Outcome: Percentage of Patients With Overall Response at Week 52
Description: Overall response after treatment at week 52 was defined as maintenance of platelet count ≥ 30 x 109/L and ≥ 2-fold increase of screening platelet count after treatment discontinuation in the absence of bleeding event ≥ Grade II and no rescue therapy at all visits until Week 52. Bleeding events ≥ Grade II are assessed by the modified World Health Organization (WHO) Bleeding Scale; Bleeding is graded based on a 1-4 scale (1=minor bleeding to 4=severe bleeding). Characteristics of bleeding events ≥ Grade II include: epistaxis ≥30 minutes, large purpura, joint bleeding, melanotic stool, hematemesis, gross hematuria, abnormal vaginal bleeding, hemoptysis, Visible blood in body cavity fluid, retinal bleeding, bleeding at invasive sites, bleeding requiring transfusion, bleeding associated with moderate or severe hemodynamic instability, fatal bleeding, CNS bleeding.
Time Frame: Study treatment discontinuation until week 52
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Participants | 2 | 2
Statistical Analysis 1: Comparison: Eltrombopag + Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.5133, Regression, Logistic

3. Secondary Outcome: Duration of Sustained Response Off Treatment
Description: Duration of sustained response off treatment is defined as time of treatment discontinuation until platelet count < 30 × 109/L or bleeding events ≥ Grade II or use of any rescue therapy. If sustained response remains, the interval was censored with the date of the last platelet assessment. Bleeding events ≥ Grade II are assessed by the modified World Health Organization (WHO) Bleeding Scale; Bleeding is graded based on a 1-4 scale (1=minor bleeding to 4=severe bleeding). Characteristics of bleeding events ≥ Grade II include: epistaxis ≥30 minutes, large purpura, joint bleeding, melanotic stool, hematemesis, gross hematuria, abnormal vaginal bleeding, hemoptysis, Visible blood in body cavity fluid, retinal bleeding, bleeding at invasive sites, bleeding requiring transfusion, bleeding associated with moderate or severe hemodynamic instability, fatal bleeding, CNS bleeding.
Time Frame: from last dose of study treatment until loss of response, approx. 52 weeks
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization and who had a response.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 2 | 2
Weeks | 49.1 (0.0) | 45.7 (2.8)

4. Secondary Outcome: Overall Response by Week 4
Description: Overall response by week 4 is defined as platelet count ≥ 30 × 109/L and ≥ 2 fold increase of screening platelet count and absence of bleeding and no rescue therapy within the first 4 weeks
Time Frame: By Week 4
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Participants | 10 | 11

5. Secondary Outcome: Complete Response by Week 4
Description: Complete Response by week 4 is defined as platelet count ≥ 100 × 109/L and absence of bleeding and no rescue therapy until week 4.
Time Frame: By Week 4
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Participants | 8 | 9

6. Secondary Outcome: Absolute Change in Platelet Count From Pre-treatment/Screening to Baseline and to Various Time Points
Description: Absolute change in platelet count from pre-treatment or screening to baseline (week 1) and from pre-treatment / screening to 2, 4, 13, 27 and 53 weeks. If pre-treatment was necessary before inclusion, platelet count data performed directly before pre-treatment were used for study inclusion (screening value to be used for inclusion/exclusion check and for analysis as a covariate).
Time Frame: Pre-treatment/screening, Week 1 (baseline), 2, 4, 13, 27, and 53
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization. Only patients who contributed data were included in the "number analyzed" per week. As not all participants contributed data for each visit the "overall number of participants analyzed" and the "number analyzed" per week differ.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 12 | 13
G/L
  Week 1: number analyzed (Participants) | 11 | 11
  Week 1 | 32.0 (44.3) | 23.2 (48.0)
  Week 2: number analyzed (Participants) | 11 | 12
  Week 2 | 145.2 (151.9) | 80.7 (68.8)
  Week 4: number analyzed (Participants) | 11 | 12
  Week 4 | 192.5 (165.8) | 92.0 (68.7)
  Week 13: number analyzed (Participants) | 10 | 11
  Week 13 | 119.4 (115.9) | 143.0 (88.5)
  Week 27: number analyzed (Participants) | 9 | 11
  Week 27 | 217.8 (126.5) | 141.2 (94.7)
  Week 53: number analyzed (Participants) | 8 | 10
  Week 53 | 139.0 (88.0) | 141.7 (61.4)

7. Secondary Outcome: Relative Change in Platelet Count From Pre-treatment/Screening to Baseline and to Various Time Points
Description: Relative change in platelet count from pre-treatment or screening to baseline (week 1) and from pre-treatment or screening to 2, 4, 13, 27, and 53 weeks. If pre-treatment was necessary before inclusion, platelet count data performed directly before pre-treatment were used for study inclusion (screening value to be used for inclusion/exclusion check and for analysis as a covariate).
Time Frame: Pre-treatment/screening, Week 1 (baseline), 2, 4, 13, 27, and 53
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage change in platelet counts
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 12 | 13
Percentage change in platelet counts
  Week 1: number analyzed (Participants) | 10 | 11
  Week 1 | 347.9 (486.8) | 293.4 (418.4)
  Week 2: number analyzed (Participants) | 10 | 12
  Week 2 | 5795.5 (9672.4) | 2028.2 (4382.0)
  Week 4: number analyzed (Participants) | 10 | 12
  Week 4 | 11400.9 (16875.2) | 2865.4 (3805.4)
  Week 13: number analyzed (Participants) | 9 | 11
  Week 13 | 8050.6 (12277.8) | 4725.7 (8418.2)
  Week 27: number analyzed (Participants) | 8 | 11
  Week 27 | 13667.9 (15717.1) | 4381.1 (8195.2)
  Week 53: number analyzed (Participants) | 7 | 10
  Week 53 | 9392.3 (11476.0) | 5612.1 (8300.7)

8. Secondary Outcome: Time to Overall Response (TOR)
Description: Time to overall response is defined as time from starting study treatment to time of achievement of overall response. Overall response is defined as a platelet count ≥ 30 × 10^9/L and ≥ 2 fold increase of baseline platelet count and absence of bleeding and no rescue therapy censored with the last visit date for patients not achieving overall response. Results of TOR are reported per Kaplan-Meier estimates.
Time Frame: Time from starting study treatment to achievement of complete response (up to 52 weeks)
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Weeks | 1.1 [0.0 to 4.1] | 1.0 [0.1 to 1.3]

9. Secondary Outcome: Time to Complete Response
Description: Time to complete response is defined as time from starting study treatment to time of achievement of complete response. Complete response is defined as a platelet count ≥ 100 × 109/L and absence of bleeding and no rescue therapy. Results of time to complete response are reported per Kaplan-Meier estimates.
Time Frame: Time from starting study treatment to achievement of complete response (up to 52 weeks)
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Weeks | 1.1 [0.1 to NA] — NA = upper limit of CI is inestimable because there were not enough events to calculate | 2.1 [0.6 to NA] — NA = upper limit of CI is inestimable because there were not enough events to calculate

10. Secondary Outcome: Duration of Overall Response (OR) and Complete Response (CR)
Description: Duration of overall or complete response (CR) is defined as time of achievement of overall or CR until loss of overall or CR. The duration of CR was calculated from the date of onset of CR until platelet count < 100 x 109/L, or bleeding events ≥ Grade II (assessed by the modified World Health Organization (WHO) Bleeding Scale) or use of any rescue therapy, whatever was earlier. Bleeding is graded based on a 1-4 scale (1=minor bleeding to 4=severe bleeding). Characteristics of bleeding events ≥ Grade II include: epistaxis ≥30 minutes, large purpura, joint bleeding, melanotic stool, hematemesis, gross hematuria, abnormal vaginal bleeding, hemoptysis, Visible blood in body cavity fluid, retinal bleeding, bleeding at invasive sites, bleeding requiring transfusion, bleeding associated with moderate or severe hemodynamic instability, fatal bleeding, CNS bleeding. Results of duration of overall and complete response are reported per Kaplan-Meier estimates.
Time Frame: Achievement of overall or complete response until loss of response (up to 52 weeks)
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization. Patients who did not reach OR/CR were censored at time 0.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Weeks
  Median duration of overall response | 8.3 [0.3 to NA] — NA = upper limit of CI is inestimable because there were not enough events to calculate | 3.6 [1.1 to NA] — NA = upper limit of CI is inestimable because there were not enough events to calculate
  Median duration of complete response | 9.7 [1.3 to NA] — NA = upper limit of CI is inestimable because there were not enough events to calculate | 1.3 [0.9 to 6.1]

11. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Questionnaire
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) instrument is a 13-item validated tool used to measure an individual's level of fatigue during usual daily activities over the past 7 days. Items are scored on a 0-4 response scale (4=not at all to 0=very much) where the total possible score ranges from 0-52 (all items are summed up to create the total score); A score of less than 30 indicates severe fatigue. The higher scores represent better HRQoL.
Time Frame: Baseline (Week 1), Week 2, 3, 5, 13, 27 and 53
Population: as for outcome 6
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 10 | 11
scores on a scale
  Change from Baseline (BL) to Week 2 | -4.2 (9.6) | -4.5 (6.9)
  Change from BL to Week: number analyzed (Participants) | 9 | 10
  Change from BL to Week | 1.0 (4.4) | -2.9 (5.1)
  Change from BL to Week 5: number analyzed (Participants) | 10 | 10
  Change from BL to Week 5 | 1.2 (5.0) | -5.1 (6.9)
  Change from BL to Week 13: number analyzed (Participants) | 8 | 9
  Change from BL to Week 13 | 0.3 (8.3) | 0.3 (2.8)
  Change from BL to Week 27: number analyzed (Participants) | 8 | 10
  Change from BL to Week 27 | -3.6 (11.0) | -3.1 (7.7)
  Change from BL to Week 53: number analyzed (Participants) | 6 | 9
  Change from BL to Week 53 | 2.7 (5.6) | -3.4 (5.4)

12. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire (Physical (PS), Mental Score (MS) and Alternative Scoring (PS-QM))
Description: SF36 questionnaire is a tool to measure health-related QoL. SF36 questionnaires (physical and mental score) were answered throughout the study and is a validated instrument with 36 questions to measure general physical and mental health status via assessment of 8 domains-Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health-over the past 4 weeks. The SF36 is scored using norm-based scoring procedures and scores ranging from 0-100; higher values indicate less impairment, a higher QoL. In addition to this SAP-planned scoring score, an alternative scoring for both the physical SF36 score and the mental SF36 were performed by QualityMetric (QM) Incorporated, an IQVIA business.
Time Frame: Baseline (Week 1), Week 2, 3, 5, 13, 27 and 53
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 11 | 12
scores on a scale
  Change from Baseline (CBL) to Wk 2: Physical Score (PS): number analyzed (Participants) | 10 | 11
  Change from Baseline (CBL) to Wk 2: Physical Score (PS) | 1.9 (4.6) | -3.3 (6.6)
  CBL to Week 3: PS: number analyzed (Participants) | 8 | 10
  CBL to Week 3: PS | 2.5 (5.8) | -1.4 (8.8)
  CBL to Week 5: PS: number analyzed (Participants) | 8 | 9
  CBL to Week 5: PS | 1.5 (6.2) | -2.7 (10.5)
  CBL to Week 13: PS: number analyzed (Participants) | 7 | 10
  CBL to Week 13: PS | 3.5 (9.9) | 0.3 (8.0)
  CBL to Week 27: PS: number analyzed (Participants) | 7 | 10
  CBL to Week 27: PS | 2.6 (14.7) | -0.9 (10.8)
  CBL to Week 53: PS: number analyzed (Participants) | 6 | 10
  CBL to Week 53: PS | 8.1 (11.8) | 0.3 (10.0)
  CBL to Week 2: Mental Score (MS): number analyzed (Participants) | 10 | 11
  CBL to Week 2: Mental Score (MS) | -0.8 (6.1) | -1.2 (7.6)
  CBL to Week 3: MS: number analyzed (Participants) | 8 | 10
  CBL to Week 3: MS | -2.0 (11.0) | -1.6 (9.7)
  CBL to Week 5: MS: number analyzed (Participants) | 8 | 9
  CBL to Week 5: MS | 0.1 (7.3) | -1.7 (11.5)
  CBL to Week 13: MS: number analyzed (Participants) | 7 | 10
  CBL to Week 13: MS | 3.3 (7.5) | 4.1 (7.4)
  CBL to Week 27: MS: number analyzed (Participants) | 7 | 10
  CBL to Week 27: MS | -1.4 (4.9) | -2.7 (7.4)
  CBL to Week 53: MS: number analyzed (Participants) | 6 | 10
  CBL to Week 53: MS | 2.1 (8.8) | 0.6 (5.7)
  CBL to Week 2: PS-QM | 2.0 (4.1) | -3.3 (6.0)
  CBL to Week 3: PS-QM: number analyzed (Participants) | 11 | 11
  CBL to Week 3: PS-QM | 3.4 (6.4) | -1.4 (7.8)
  CBL to Week 5: PS-QM: number analyzed (Participants) | 9 | 12
  CBL to Week 5: PS-QM | 2.4 (6.0) | -2.7 (8.5)
  CBL to Week 1: PS-QM: number analyzed (Participants) | 10 | 10
  CBL to Week 1: PS-QM | 4.1 (8.5) | 0.3 (7.6)
  CBL to Week 27: PS-QM: number analyzed (Participants) | 9 | 11
  CBL to Week 27: PS-QM | 3.6 (12.4) | -1.0 (9.7)
  CBL to Week 53: PS-QM: number analyzed (Participants) | 7 | 10
  CBL to Week 53: PS-QM | 6.2 (10.7) | 0.2 (9.4)

13. Secondary Outcome: Incidence and Severity of Bleeding Events
Description: Incidence and severity of bleeding assessed by the modified World Health Organization (WHO) Bleeding Scale; Bleeding is graded based on a 1-4 scale (1=minor bleeding to 4=severe bleeding).
  Incidence of bleeding: participants had at least one bleeding event. Severity of bleeding: bleeding event is from grade 2 and higher
Time Frame: Baseline up to 52 weeks
Population: The Full Analysis Set (FAS) consists of all patients to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
Number analyzed (Participants) | 13 | 13
Participants
  Incidence of Bleeding events | 10 | 12
  Incidence of Bleeding events with severity: ≥ grade 2 | 6 | 2
  Incidence of Bleeding events with severity: ≥ grade 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are collected from the first dose of study treatment until end of study treatment plus 30 days post treatment for each patient. AEs reported in this record are from first dose of study treatment until 30 days after end of treatment for each patient, approx. 3 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Arm/Group | Eltrombopag + Dexamethasone | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/13
Serious Adverse Events (participants affected / at risk) | 5/12 | 5/13
Other Adverse Events (participants affected / at risk) | 11/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag + Dexamethasone (N=12) | Dexamethasone (N=13)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag + Dexamethasone (N=12) | Dexamethasone (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 3
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 4
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 3 | 4
Gastroenteritis viral (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Keratitis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Nervousness (Psychiatric disorders) | 1 | 0
Nocturnal fear (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04346654/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04346654/SAP_001.pdf